CLINICAL TRIAL: NCT03357120
Title: Detection of Circulating Tumoral DNA Mutations (Sequential Assessment) Following Neoadjuvant Chemotherapy for Breast Cancer: Clinical Validity (ALIENOR Study)
Brief Title: Circulating Tumor DNA After Neoadjuvant Chemotherapy
Acronym: ALIENOR
Status: Recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: Institut Bergonié (Other)
Collaborators: Fondation Bergonié (Unknown)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Other
Other Study IDs: IB 2017-02; ID-RCB number : 2017-A00939-44 (Other: ANSM)
Record Dates: First submitted 2017-11-09; First posted 2017-11-29 (Actual); Last update posted 2025-10-02 (Actual); Status verified 2025-10

CONDITIONS: Breast Cancer
Keywords: Breast Cancer; Neoadjuvant chemotherapy; Circulating tumor DNA
MeSH Terms: conditions — Breast Neoplasms

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (1):
- Follow-up after neoadjuvant chemotherapy (Other): Patients with an invasive breast cancer on neoadjuvant chemotherapy (with the exception of cT2cN0 tumors) are preselected before the surgical procedure. They are definitely included during the post-surgery visit following the analysis of the surgical specimen (only patients whose tumor did not achieve a complete pathological response are included).
  Interventions: Other: Follow-up after neoadjuvant chemotherapy

INTERVENTIONS:
Other: Follow-up after neoadjuvant chemotherapy — Sequential plasma samples for ctDNA mutations analysis will be taken during the post-surgery visit (within 2-5 weeks after surgery) and every 6 months (+/- 1 month) thereafter for 5 years. In case of relapse patients will be proposed to participate to an optional research program with a blood test for ctDNA assessment and biopsies from a metastasis (when these biopsies are clinically indicated). Next Generation Sequencing (NGS) analysis will be performed on post-neoadjuvant chemotherapy residual tumor tissue samples. The mutations identified by NGS in residual tumor will be tracked in ctDNA using personalized digital PCR (dPCR) or by an NGS technique whose bioinformatics pipeline is adapted to the analysis of ctDNA.
  In case of relapse patients will be proposed to participate to an optional research program with a blood test for ctDNA assessment and biopsies from a metastasis (when these biopsies are clinically indicated).

SUMMARY:
Trial assessing the prognostic value of ctDNA mutations from samples taken sequentially in patients with invasive breast cancer initially treated with neoadjuvant chemotherapy and whose tumor is not in complete histological response.

DETAILED DESCRIPTION:
Patients with an invasive breast cancer on neoadjuvant chemotherapy (with the exception of cT2cN0 tumors) are preselected before the surgical procedure. They are definitely included during the post-surgery visit following the analysis of the surgical specimen (only patients whose tumor did not achieve a complete pathological response are included).

Sequential plasma samples for ctDNA mutations analysis will be taken during the post-surgery visit (within 2-5 weeks after surgery) and every 6 months (+/- 1 month) thereafter for 5 years.

In case of relapse patients will be proposed to participate to an optional research program with a blood test for ctDNA assessment and biopsies from a metastasis (when these biopsies are clinically indicated).

ELIGIBILITY:
Inclusion Criteria :

1. Age ≥ 18 years (no age limit).
2. Women or men.
3. Invasive breast cancer proven histologically at diagnosis (before neoadjuvant chemotherapy):

   1. Locally advanced tumor known to be inoperable from the start:

      * cT4a, b, c, d whatever the cN
      * or cN2 or cN3 whatever the cT.
   2. Operable tumors:

      * cT2cN1 or cT3cN0 or cT3N1,
      * or cT2cN0 for which ganglionic invasion has been proven by cytology or histology.
4. Lack of clinically or radiologically detectable metastases in the initial diagnosis before the neoadjuvant chemotherapy (M0).
5. Unilateral or bilateral breast cancer. Multifocality is accepted.
6. Patients who received 6 to 8 cycles of neoadjuvant chemotherapy.
7. Preoperative radiation therapy allowed.
8. Breast surgery performed and pathology report of a non-complete histological response (i.e. all the different results of ypT0 /is ypN0).
9. Signed informed consent.
10. Patients affiliated to a French social security scheme in accordance with Article 1121-11 of the French Code of Public Health.
11. Possible inclusion in another interventional research (surgical, radiotherapy or drug study).

Exclusion Criteria :

1. cT2cN0 tumor without cytological or histological lymph node involvement.
2. Progression during neoadjuvant chemotherapy.
3. Exclusive neoadjuvant hormone therapy.
4. Complete blood transfusion within 120 days prior to 1st sampling.
5. History of invasive cancer regardless of the time elapsed since the diagnosis of this cancer, including a history of contralateral invasive breast cancer. However, patients who have been treated for in situ breast cancer, basocellular skin cancer or cervical cancer treated in situ are eligible.
6. Patient unable to follow and comply with research procedures for geographical, social or psychological reasons.
7. Patient deprived of liberty or subject to a legal protection measure.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 180 (Estimated)
Dates: Start 2017-10-06 (Actual); Primary Completion 2026-10 (Estimated); Study Completion 2028-10 (Estimated)

PRIMARY OUTCOMES:
Prognostic value of the presence of ctDNA mutation(s) measured by dPCR on recurrence-free interval (RFI) at 3 years. | 3 years

SECONDARY OUTCOMES:
Prognostic value of the presence of ctDNA mutation(s) on overall survival (OS) at 3 years. | 3 years
Prognostic value of the presence of ctDNA mutation(s) on distant-metastasis-free interval (DRFI) at 3 years. | 3 years
Prognostic value of the presence of ctDNA mutation(s) on OS at 5 years. | 5 years
Prognostic value of the presence of ctDNA mutation(s) on DRFI at 5 years. | 5 years
Prognostic value of the presence of ctDNA mutation(s) on a single sample assessment after surgery (measured by dPCR) on RFI at 3 years. | 3 years
Prognostic value of the presence of ctDNA mutation(s) on a single sample assessment after surgery (measured by dPCR) on DRFI at 3 years. | 3 years
Prognostic value of the presence of ctDNA mutation(s) on a single sample assessment after surgery (measured by dPCR) on RFI at 5 years. | 5 years
Prognostic value of the presence of ctDNA mutation(s) on a single sample assessment after surgery (measured by dPCR) on DRFIat 5 years. | 5 years

CONTACTS AND LOCATIONS:
Overall Officials: Hervé BONNEFOI, MD, PhD, Study Chair — Institut Bergonié
Locations (1):
- Institut Bergonie, Bordeaux, France

IPD SHARING:
Plan to Share IPD: No